CLINICAL TRIAL: NCT01832753
Title: Levothyroxine Treatment and Cardiometabolic Outcomes in Adolescents With Down Syndrome
Brief Title: Treatment Trial of Subclinical Hypothyroidism in Down Syndrome
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Children's Hospital of Philadelphia (Other)
Collaborators: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 12-009578; 1R01HD071981-01A1 (NIH)
Record Dates: First submitted 2013-04-09; First posted 2013-04-16 (Estimated); Results first posted 2019-06-13 (Actual); Last update posted 2019-09-06 (Actual); Status verified 2019-09

CONDITIONS: Down Syndrome; Subclinical Hypothyroidism
Keywords: Down syndrome; subclinical hypothyroidism; thyroid; levothyroxine
MeSH Terms: conditions — Down Syndrome; Thyroid Diseases | interventions — Thyroxine

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Treatment Phase: Months 6-18 (Placebo Comparator): Subject who are found to have SCH at the 6-month visit will be randomized to receive either levothyroxine or placebo during months 6-12. Levothyroxine dose will be between 0.5 - 1 mcg/kg/day. There will be 1 blood draw visit at month 7.5 (6 weeks after randomization) and 1 study visit at month 12 that will provide the opportunity for dose adjustments if needed.
  From months 12-18, all subjects will receive levothyroxine. Levothyroxine dose will be between 0.5 - 1 mcg/kg/day. There will be one blood draw visit at month 13.5 that will provide the opportunity for dose adjustments if needed.
  Interventions: Drug: Levothyroxine
- Observation Phase: Months 0-6 (No Intervention): Subjects will be observed for the first 6 months of the study to ensure that the subclinical hypothyroidism is persistent. Subjects who do not have SCH at 6 months will not proceed to the treatment phase.
  Subjects that have TSH >10 mIU/L during the 6 month Observational Phase will not be considered subclinical and will not qualify to continue the study. They will be referred to an endocrinologist for treatment.

INTERVENTIONS:
Drug: Levothyroxine
  Other Names: Synthroid; Levothroid; Levoxyl; Tirosint; Unithroid
  Arms: Treatment Phase: Months 6-18

SUMMARY:
The purpose of this research study is to learn about the effects of treating subclinical hypothyroidism (SCH) with thyroid hormone replacement in children and adolescents with Down syndrome (DS). We hypothesize that treatment of SCH with thyroid hormone replacement will improve cardiometabolic health and quality of life.

DETAILED DESCRIPTION:
The American Academy of Pediatrics (AAP) recommends yearly screening of thyroid studies in DS. Clinical experience suggests that thyroid stimulating hormone (TSH) concentrations in the subclinical hypothyroid range (5-10 milli international units(mIU/L)) are not uncommon in DS, but the benefits and risks of treating SCH in the DS population are not known. In adults, SCH has been associated with increased cardiometabolic risk (CMR) and individuals with DS may be at increased cardiometabolic risk as well.

Data in children with SCH are limited. Despite the recommendations to screen for thyroid dysfunction, evidence to guide management of elevated TSH in children with DS is equally sparse. In non-DS children, TSH>4.65 mIU/L was associated with lower HDL. One year of levothyroxine treatment in short children with subclinical hypothyroidism and short stature improved growth velocity. Left ventricular (LV) function and LV mass (by echocardiography) was not different in 16 children with DS and subclinical hypothyroidism (TSH>6.5 mIU/L; mean TSH = 7.8 mIU/L) vs. 25 children with DS and normal TSH. However, these findings may be limited by the small sample size. An intervention study of 7 subjects age 2-42 years with DS and hypothyroidism, defined as low T4 and normal or elevated TSH (0.2-18.9 mIU/L) on 8 weeks of levothyroxine treatment did not improve developmental or functional outcomes. Anthropometrics and CMR factors were not examined. In contrast, increased TSH in the absence of overt congenital hypothyroidism is common in neonates with DS and prompted a randomized controlled trial (RCT) in 181 neonates with DS. TSH-directed levothyroxine treatment was associated with better growth, weight gain, and motor development after 24 months compared to placebo. These findings highlight that the "asymptomatic" component of subclinical hypothyroidism may have medically-relevant effects. This study will provide potentially clinically relevant preliminary evidence for the treatment of subclinical hypothyroidism in DS.

ELIGIBILITY:
Inclusion Criteria:

* Males and females, ages 8 - 20 years
* Diagnosis of Down syndrome
* Subclinical hypothyroidism: TSH level between 5 - 10 mIU/L, normal T4
* Parental/guardian permission (informed consent) and if appropriate, child assent
* Females who are at least 11 years of age or who are menarchal must have a negative urine/serum pregnancy test
* Committed to adherence to levothyroxine treatment and study completion

Exclusion Criteria:

* Pregnancy
* Type 1/Type 2 diabetes
* Chronic medical conditions or medication use that can affect growth, nutrition, blood glucose, insulin secretion, or thyroid function (such as lithium or certain seizure medications)
* Current use of levothyroxine or anti-thyroid hormone
* Cyanotic congenital heart disease, or pulmonary hypertension (as described by last echo report in subjects with CHD), or congenital heart disease considered medically unstable by the study cardiologists

Ages: 8 Years to 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 12 (Actual)
Dates: Start 2013-01 (Actual); Primary Completion 2017-10-18 (Actual); Study Completion 2017-10-18 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Andrea Kelly, MD, MSCE, Principal Investigator — Children's Hospital of Philadelphia
Locations (2):
- United States (2):
  - Children's National Medical Center, Washington D.C., District of Columbia
  - The Children's Hospital of Philadelphia, Philadelphia, Pennsylvania

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Immediate Treatment: Subjects in this group were observed during months 0-6, were randomized to receive levothyroxine during months 6-12, and received levothyroxine as part of the open label phase months 12-18.
  All doses were between between 0.5 - 1 mcg/kg/day.
- Delayed Treatment: Subjects in this group were observed during months 0-6, were randomized to receive placebo during months 6-12, and received levothyroxine as part of the open label phase months 12-18.
  All doses were between between 0.5 - 1 mcg/kg/day.
- Observation Only: Subjects in this group partook in the study during the observational phase months 0-6. Subjects in this group were not randomized to either immediate or delayed treatment groups.
Period: Observation Phase (Months 0-6)
Arm/Group | Immediate Treatment | Delayed Treatment | Observation Only
Started | 5 | 4 | 3
Completed | 5 | 4 | 1
Not Completed | 0 | 0 | 2
Period: Randomization Phase (Months 6-12)
Arm/Group | Immediate Treatment | Delayed Treatment | Observation Only
Started | 5 | 4 | 0 (1 subject was not randomized as they did not meet inclusion criteria at the end of observation phase)
Completed | 4 | 3 | 0
Not Completed | 1 | 1 | 0
Period: Open Label Dose Phase (Months 12-18)
Arm/Group | Immediate Treatment | Delayed Treatment | Observation Only
Started | 3 | 3 | 0
Completed | 3 | 3 | 0
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Immediate Treatment | Delayed Treatment | Observation Only | Total
Number analyzed (Participants) | 5 | 4 | 3 | 12
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 12.4 [9.9 to 15.2] | 11.6 [8.7 to 14.4] | 16.5 [14.7 to 18.6] | 14.0 [10.2 to 15.8]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 4 | 2 | 10
  Male | 1 | 0 | 1 | 2
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 0 | 0 | 1
  Not Hispanic or Latino | 4 | 4 | 3 | 11
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 1 | 2 | 0 | 3
  White | 3 | 2 | 3 | 8
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 1 | 0 | 0 | 1
Region of Enrollment [Number; unit: participants]
  United States | 5 | 4 | 3 | 12
BMI Percentile [Median (Inter-Quartile Range); unit: Percentile] | 94 [76 to 99] | 98 [77 to 99] | 98 [76 to 99] | 98 [76 to 99]

OUTCOME MEASURES:

1. Primary Outcome: Change in Lipid Panel From Baseline at 6, 12 and 18 Months.
Description: Lipid panel will be measured via fasting blood draw.
Time Frame: baseline, 6 months, 12 months & 18 months
Population: 3 of the 12 participants ("Observation Only") were withdrawn prior to randomization due to normal TSH. 1 of the 4 Delayed Treatment group participants self-withdrew before their 12 month visit. 1 of the 5 Immediate Treatment participants withdrew due to elevated TSH at their 12 month visit, 1 and self-withdrew before their 12 month visit.
Measure: Median (Inter-Quartile Range); unit: mg/dL
Arm/Group | Immediate Treatment | Delayed Treatment | Observation Only
Number analyzed (Participants) | 5 | 4 | 3
mg/dL
  Baseline Cholesterol (mg/dL) | 160 [145 to 208] | 170 [144 to 201] | 163 [150 to 201]
  6 month Cholesterol (mg/dL): number analyzed (Participants) | 5 | 4 | 1
  6 month Cholesterol (mg/dL) | 172 [159 to 203] | 156.5 [133 to 203.5] | 226 [226 to 226]
  12 month Cholesterol (mg/dL): number analyzed (Participants) | 4 | 3 | 0
  12 month Cholesterol (mg/dL) | 178.5 [147.5 to 215] | 172 [149 to 191] |
  18 month Cholesterol (mg/dL): number analyzed (Participants) | 3 | 3 | 0
  18 month Cholesterol (mg/dL) | 150 [150 to 217] | 164 [134 to 214] |
  Baseline HDL-C (mg/dL) | 44 [38 to 46] | 45.5 [40 to 49.5] | 43 [32 to 47]
  6 month HDL-C (mg/dL): number analyzed (Participants) | 5 | 4 | 1
  6 month HDL-C (mg/dL) | 35 [32 to 40] | 46.5 [42.5 to 50] | 48 [48 to 48]
  12 month HDL-C (mg/dL): number analyzed (Participants) | 4 | 3 | 0
  12 month HDL-C (mg/dL) | 42.5 [40.5 to 43] | 44 [37 to 50] |
  18 month HDL-C (mg/dL): number analyzed (Participants) | 3 | 3 | 0
  18 month HDL-C (mg/dL) | 38 [36 to 42] | 47 [43 to 49] |
  Baseline LDL-C (mg/dL) | 101 [91 to 145] | 108 [82.5 to 133.5] | 95 [89 to 138]
  6 month LDL-C (mg/dL): number analyzed (Participants) | 5 | 4 | 1
  6 month LDL-C (mg/dL) | 117 [116 to 120] | 96.5 [74.5 to 134.5] | 161 [161 to 161]
  12 month LDL-C (mg/dL): number analyzed (Participants) | 4 | 3 | 0
  12 month LDL-C (mg/dL) | 111 [88 to 139.5] | 101 [96 to 133] |
  18 month LDL-C (mg/dL): number analyzed (Participants) | 3 | 3 | 0
  18 month LDL-C (mg/dL) | 90 [90 to 104] | 99 [79 to 148] |
  Baseline nonHDL-C (mg/dL) | 116 [108 to 160] | 124.5 [94.5 to 161] | 118 [116 to 158]
  6 month nonHDL-C (mg/dL): number analyzed (Participants) | 5 | 4 | 1
  6 month nonHDL-C (mg/dL) | 134 [132 to 160] | 108 [87 to 157] | 178 [178 to 178]
  12 month nonHDL-C (mg/dL): number analyzed (Participants) | 4 | 3 | 0
  12 month nonHDL-C (mg/dL) | 137.5 [107 to 172] | 122 [105 to 154] |
  18 month nonHDL-C (mg/dL): number analyzed (Participants) | 3 | 3 | 0
  18 month nonHDL-C (mg/dL) | 112 [108 to 181] | 115 [87 to 171] |
  Basline Triglycerides (mg/dL) | 73 [73 to 84] | 88 [61.5 to 137] | 117 [98 to 133]
  6 month Triglycerides (mg/dL): number analyzed (Participants) | 5 | 4 | 1
  6 month Triglycerides (mg/dL) | 91 [75 to 96] | 83 [61 to 116] | 84 [84 to 84]
  12 month Triglycerides (mg/dL): number analyzed (Participants) | 4 | 3 | 0
  12 month Triglycerides (mg/dL) | 99 [80.5 to 178] | 106 [45 to 107] |
  18 month Triglycerides (mg/dL): number analyzed (Participants) | 3 | 3 | 0
  18 month Triglycerides (mg/dL) | 108 [91 to 383] | 82 [38 to 113] |

2. Secondary Outcome: Change in Quality of Life From Baseline at 6, 12 and 18 Months.
Description: Questionnaires will be done with participants and parents on the day of each study visit to determine body image and quality of life. The Pediatric Quality of Life (PedsQL) scale is a 5-item scale (values 1-5). 1 - "Always True", to 5 - "Never True". Items are reverse-scored and linearly transformed to a 0-100 scale (0 = 100, 1 = 75, 2 = 50, 3 = 25, 4 = 0), so that greater scores indicate better QOL.
Time Frame: baseline, 6 months, 12 months, & 18 months
Population: as for outcome 1
Measure: Median (Full Range); unit: Unit on a scale, linearly transformed
Arm/Group | Immediate Treatment | Delayed Treatment | Observation Only
Number analyzed (Participants) | 5 | 4 | 3
Unit on a scale, linearly transformed
  Baseline Pediatric Quality of Life | 70.65 [59.78 to 83.7] | 69.02 [54.35 to 92.39] | 52.17 [51.09 to 57.61]
  6 month Pediatric Quality of Life: number analyzed (Participants) | 4 | 4 | 1
  6 month Pediatric Quality of Life | 66.305 [57.61 to 75] | 61.41 [54.35 to 93.48] | 50 [50 to 50]
  12 month Pediatric Quality of Life: number analyzed (Participants) | 3 | 2 | 0
  12 month Pediatric Quality of Life | 75 [64.13 to 84.78] | 76.085 [56.52 to 95.65] |
  18 month Pediatric Quality of Life: number analyzed (Participants) | 2 | 3 | 0
  18 month Pediatric Quality of Life | 70.655 [54.35 to 86.96] | 90.22 [50 to 94.57] |

ADVERSE EVENTS:
Time Frame: Adverse Events were collected throughout the course of the study at each study visit and weekly following randomization up to 18 months.
Description: Adverse Events are tracked over groups divided by phase of study for the purpose of full transparency of the relationship between study drug and AEs.
Groups:
- Observation Phase: Months 0-6
  Subjects will be observed for the first 6 months of the study to ensure that the subclinical hypothyroidism is persistent. Subjects who do not have SCH at 6 months will not proceed to the treatment phase.
  Subjects that have TSH >10 mIU/L during the 6 month Observational Phase will not be considered subclinical and will not qualify to continue the study. They will be referred to an endocrinologist for treatment.
- Randomization Phase - Placebo: Months 6-12
  This group includes those 4 out of 12 participants that were randomized to the delayed treatment group and received placebo for months 6-12. Adverse events will be reported in this column of the table if the AEs occurred during the phase in which participants were receiving placebo.
- Randomization Phase - Treatment: Months 6-12
  This group includes those 5 of 12 participants that were randomized to immediate treatment. Levothyroxine dose is between 0.5 - 1 mcg/kg/day. There is 1 blood draw visit at month 7.5 (6 weeks after randomization) and 1 study visit at month 12 that will provide the opportunity for dose adjustments if needed.
  From months 12-18, all subjects will receive levothyroxine. Levothyroxine dose will be between 0.5 - 1 mcg/kg/day. There will be one blood draw visit at month 13.5 that will provide the opportunity for dose adjustments if needed.
- Open Label Treatment Phase: Months 12-18
  6 of the starting 12 participants took part in this phase of the study; 3 from the delayed treatment aka placebo group, 3 from the immediate treatment group. From months 12-18, all subjects receive levothyroxine. Levothyroxine dose is between 0.5 - 1 mcg/kg/day. There is one blood draw visit at month 13.5 that will provide the opportunity for dose adjustments if needed.
Arm/Group | Observation Phase | Randomization Phase - Placebo | Randomization Phase - Treatment | Open Label Treatment Phase
All-Cause Mortality (participants affected / at risk) | 0/12 | 0/4 | 0/5 | 0/6
Serious Adverse Events (participants affected / at risk) | 0/12 | 0/4 | 0/5 | 0/6
Other Adverse Events (participants affected / at risk) | 1/12 | 4/4 | 4/5 | 1/6
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Observation Phase (N=12) | Randomization Phase - Placebo (N=4) | Randomization Phase - Treatment (N=5) | Open Label Treatment Phase (N=6)
Anxiety Symptoms (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) — hair pulling & difficulty urinating, unlikely related to study
Dry mouth (General disorders) | 0 (0) | 1 (3) | 0 (0) | 0 (0) — Chapped lips, dry mouth, unlikely related to study
Diarrhea (Gastrointestinal disorders) | 1 (1) | 2 (2) | 1 (1) | 0 (0) — unlikely related
Racing Heart (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) — Racing Heart, Light Headedness, possibly related
Skin irritation (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) — Rash on back, unlikely related to study, resolved without intervention
Sleeplessness (General disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) — not sleeping through the night, restless, irritable, unlikely related to study
Tired (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) — possibly related to study, followed up with TSH/T4 check

LIMITATIONS AND CAVEATS:
This was a pilot and feasibility study. The number of children with Down syndrome who had elevated TSH (5-10 IU/mL) and who were not on thyroid hormone replacement limited our ability to recruit.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2015-09-23): https://cdn.clinicaltrials.gov/large-docs/53/NCT01832753/Prot_SAP_000.pdf